Statistical Analysis Plan for Protocol E7080: Post-FDA Approval Clinical Trial Evaluating Bronchial Thermoplasty in Severe Persistent Asthma

NCT: NCT01350336

Document Date: 27 Jun 2016

THESE DOCUMENTS ARE THE PROPERTY OF BOSTON SCIENTIFIC CORP. AND SHALL NOT BE REPRODUCED, DISTRIBUTED, DISCLOSED OR USED FOR MANUFACTURE OR SALE OF APPARATUS WITHOUT THE EXPRESS WRITTEN CONSENT OF BOSTON SCIENTIFIC CORP.

# **Statistical Analysis Plan**

Post-FDA Approval Clinical Trial Evaluating Bronchial Thermoplasty in Severe Persistent
Asthma
PAS2

Study Reference Number E7080 (BSC), 10-02 (Asthmatx)

# CONFIDENTIAL DO NOT COPY OR DISTRIBUTE WITHOUT WRITTEN PERMISSION

# TABLE OF CONTENTS

| P | ROTO | COL SUMMARY | . 4 |
|---|------|---------------------------------------------|-----|
| 1 | INT | RODUCTION | . 6 |
| 2 | EN | DPOINT ANALYSIS | . 6 |
| | 2.1 | Primary Endpoint | . 6 |
| | 2.1 | 1 Hypotheses | . 6 |
| | 2.1 | 2 Sample Size | . 6 |
| | 2.1 | 3 Statistical Methods | . 7 |
| | 2.2 | Secondary Endpoints | . 8 |
| | 2.2 | 1 Hypotheses | . 9 |
| | 2.2 | | |
| 3 | GE | NERAL STATISTICAL METHODS | . 9 |
| | 3.1 | Analysis Sets | . 9 |
| | 3.2 | Control of Systematic Error/Bias | . 9 |
| | 3.3 | Number of Subjects per Investigative Site | . 9 |
| 4 | AD | DITIONAL DATA ANALYSES | . 9 |
| | 4.1 | Interim Analyses | . 9 |
| | 4.2 | Subgroup Analyses | 10 |
| | 4.3 | Justification of Pooling | 10 |
| | 4.4 | Multivariable Analyses | 10 |
| | 4.5 | Other Analyses | 10 |
| | 4.6 | Safety Analyses | 11 |
| | 4.7 | Changes to Planned Analyses | 12 |
| 5 | Val | idation | 12 |
| 6 | Pro | gramming Considerations | 13 |
| | 6.1 | Statistical Software | 13 |
| | 6.2 | Format of Output | 13 |
| | 6.3 | Methods for Handling Missing Data | 13 |
| | 6.4 | Identification of Severe Exacerbations (SE) | 13 |
| | 6.5 | Medication Dose Conversions | |
| 7 | Rev | vision History | 15 |

## PROTOCOL SUMMARY

| Objective(s) | The objective of this study is to evaluate durability of treatment effect and to continue to evaluate the short-term and longer-term safety profile of the Alair System in the United States and Canada in the intended use population (patients 18 years and older with severe persistent asthma) following FDA approval. |
|---|---|
| <b>Test Device</b> | Alair System for Bronchial Thermoplasty |
| <b>Control Device</b> | None |
| Study Design | This will be an open-label, single arm study designed to demonstrate durability of the treatment effect and to evaluate the short-term and longer-term safety profile of the Alair System in the United States and Canada in the intended use population (patients 18 years and older with severe persistent asthma). |
| Planned<br>Subjects/<br>Centers/<br>Countries | Up to 300 subjects (minimum of 250 subjects) will be enrolled to achieve at least 200 evaluable study subjects, accounting for a 20% drop-out rate over 5 years. The study will be conducted at a minimum of 15, and a maximum of 30, centers in the United States and Canada, limiting the number of subjects enrolled in Canada to no greater than 20%. |
| Primary<br>Endpoints | The primary endpoint will be the proportion of subjects experiencing severe exacerbations during the subsequent 12 month (for Years 2, 3, 4, and 5) compared to the first 12 month after the Alair treatment. |
| Patient<br>Success<br>Criteria | The primary statistical objective is to demonstrate that the proportion of subjects who experience severe exacerbations in the subsequent 12-mont follow-up (for Year 2, Year 3, Year 4 and Year 5 [in 12-month periods]) is not statistically worse when compared with the proportion of the first 12-months, which begins 6-weeks after the last Alair treatment. This objective will be met if the upper 95% confidence limit of the difference in proportions (i.e., the subsequent 12-month proportion minus the first 12-month proportion) is less than 20%. |
| Secondary<br>Endpoints | The secondary endpoints will include the following additional safety endpoints which will be evaluated annually through Year 5 following treatment with the Alair System: • Rates of Severe exacerbations (exacerbations / subject / year) • Respiratory adverse events* (rates of respiratory adverse events, and proportion of subjects with respiratory adverse events) |

| | <ul> <li>Emergency room visits for respiratory symptoms (rates of emergency room visits and proportion of subjects with emergency room visits for respiratory symptoms)</li> <li>Hospitalizations for respiratory symptoms (hospitalizations/ subject/ year and the proportion of subjects with hospitalizations for respiratory symptoms)</li> <li>Respiratory Serious Adverse Events (detailed narratives will be</li> </ul> |
|---|---|
| | provided for each event) • Pre- and post-bronchodilator FEV <sub>1</sub> * A respiratory adverse event is defined as any sign, symptom, illness, clinically significant abnormal laboratory value, or other adverse medical event associated with the "Respiratory System" that appears or worsens in a subject during a clinical study, regardless of whether or not it is considered related to the procedure used as part of the protocol. |
| Follow-up<br>Schedule | A follow-up evaluation will be conducted at 6 weeks after the last treatment session. At this time, the 5 year follow-up phase will begin. Subjects will be contacted via phone every 3 months to solicit for adverse events and asthma status. An in-office follow-up evaluation will be performed annually starting after the 6 week evaluation. |
| Study<br>Duration | Subjects treated with the Alair System will be followed for 5 years after the final procedure. |

#### 1 INTRODUCTION

This statistical plan addresses the planned analyses for the PAS2 Trial based on the protocol # 90889079. Specified analyses may be used for scientific presentations and/or manuscripts and may not all be provided to Regulatory Authorities.

#### 2 ENDPOINT ANALYSIS

#### 2.1 Primary Endpoint

The primary endpoint will be the proportion of subjects experiencing severe exacerbations during the subsequent 12-month period (for Years 2, 3, 4, and 5) compared to the first 12-month period after the Alair treatment.

Note: Severe exacerbation is defined as worsening of asthma symptoms requiring use of systemic corticosteroids (tablets, suspension, or injection). For subjects already taking oral corticosteroids on a daily or alternate day basis, a severe exacerbation will be defined as a worsening of asthma symptoms requiring any increase in daily dose of systemic corticosteroids. For consistency, courses of corticosteroids separated by 1 week or more will be treated as separate severe exacerbations.

The primary statistical objective is to demonstrate that the proportion of subjects who experience severe exacerbations in the subsequent 12-month follow-up (for Year 2, Year 3, Year 4 and Year 5 [in 12-month periods]) is not statistically worse when compared with the proportion of the first 12-months, which begins 6 weeks after the last Alair treatment. This objective will be met if the upper 95% confidence limit of the difference in proportions (i.e., the subsequent 12-month proportion minus the first 12-month proportion) is less than 20%.

#### 2.1.1 Hypotheses

The null and alternative hypotheses for the primary endpoint are as follows:

$$H_o: p_k - p_1 \ge 20\%$$

$$H_a: p_k - p_1 < 20\%$$

where  $p_1$  is the proportion of patients with severe exacerbations at 1 year,  $p_k$  is the proportion of patients with severe exacerbations at k years and k = 2, 3, 4, or 5.

#### 2.1.2 Sample Size

Under the assumption that in the population of US subjects treated with the Alair System the proportion of patients that experience severe exacerbations will be 0.33 (33% of subjects) or less (based on data from AIR2 Trial - 30.9%, 95% CI 24.2%, 37.7%), a sample size of 200 is adequate to demonstrate durability of the treatment effect at 5 years post-Alair treatment. Up to 300 subjects (minimum of 250 subjects) will be enrolled to achieve at least 200 evaluable study subjects, accounting for a 20% drop-out rate over 5 years. To be counted as an evaluable subject, a subject must have either completed the 5-year visit no earlier than the start of the visit

window (1797 days) or have at least 1797 days of study follow-up (see Section 2.1.3) and have primary endpoint data at 5 years.

nQuery Advisor Version 7.0 was used to form a basis for the sample size estimation. The "Two group test of equivalence in proportions (large unequal n's)" procedure based on a one-sided test at alpha equal to 0.05 and a 20% delta was used to generate the powers presented in Table 1. A minimum of 80% power was achieved for all situations wherein the subsequent year's assumed proportion of subjects with severe exacerbations was 41% or less. The use of independent samples methodology provides a conservative (over-powered) sample size calculation for matched data on a single sample.

**Table 1.** Two group test of equivalence in proportions (large unequal n's) [from nQuery Advisor 7.0]

| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
|---|---|---|---|---|---|---|---|---|---|
| Test significance level, α (one-sided) | 0.050 | 0.050 | 0.050 | 0.050 | 0.050 | 0.050 | 0.050 | 0.050 | 0.050 |
| Standard proportion, $\pi_S$ | 0.330 | 0.330 | 0.330 | 0.330 | 0.330 | 0.330 | 0.330 | 0.330 | 0.330 |
| Equivalence limit difference, $\pi_T$ - $\pi_S$ , $\Delta_0$ | 0.200 | 0.200 | 0.200 | 0.200 | 0.200 | 0.200 | 0.200 | 0.200 | 0.200 |
| Test expected proportion, $\pi_T$ | 0.330 | 0.340 | 0.350 | 0.360 | 0.370 | 0.380 | 0.390 | 0.400 | 0.410 |
| Expected difference, $\pi_T$ - $\pi_S$ , $\Delta_1$ | 0.000 | 0.010 | 0.020 | 0.030 | 0.040 | 0.050 | 0.060 | 0.070 | 0.080 |
| Power (%) | 99 | 99 | 99 | 98 | 97 | 95 | 92 | 88 | 83 |
| $n_{\rm s}$ | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 | 250 |
| $n_{\mathrm{T}}$ | 200 | 200 | 200 | 200 | 200 | 200 | 200 | 200 | 200 |
| Ratio: n <sub>T</sub> / n <sub>s</sub> | 0.800 | 0.800 | 0.800 | 0.800 | 0.800 | 0.800 | 0.800 | 0.800 | 0.800 |
| $N = n_s + n_T$ | 450 | 450 | 450 | 450 | 450 | 450 | 450 | 450 | 450 |

#### 2.1.3 Statistical Methods

See Section 6.4 for how to identify severe exacerbations.

The proportions of patients with severe exacerbations at each year  $(p_k, k=1 \text{ to } 5)$  will be calculated in two ways:

- 1. <u>Complete Follow-up:</u> using patients who complete the annual follow-up visit or have a follow-up visit (office or phone call) after the visit for that particular year if the annual visit is missed.
- 2. <u>Complete/Partial Follow-up</u>: using patients who complete the annual follow-up visit no earlier than the start of the follow-up window, have a follow-up visit (office or phone call) after the visit for that particular year if the annual visit is missed, have sufficient follow-up for the year, or had a severe exacerbation during the time period regardless of the amount of follow-up. Sufficient follow-up is having any follow-up visit (office or phone call), adverse event onset date, or hospitalization date that gives the patient at least the number of days of follow-up after the last BT procedure + 42 days given in Table 2.

Table 2. Days for sufficient follow-up by follow-up time

| Time | Days for sufficient follow-up after the follow-up period starts* |
|---|---|
| 1 Year | 337 days |
| 2 Years | 702 days |
| 3 Years | 1067 days |
| 4 Years | 1432 days |
| 5 Years | 1797 days |

<sup>\* -</sup> the follow-up period starts at last BT procedure + 42 days. The number of days in this column represents the start of the follow-up window after the follow-up period starts and is calculated as # years times 365 days minus 28 days.

All analyses will be done for patients with Complete and Complete/Partial Follow-up. Point estimates and 95% confidence intervals for the proportion of subjects experiencing severe exacerbations during each of the 12-month evaluation periods will be provided. Additionally, the exact upper 95% confidence limit for the difference between the subsequent 12-month proportions and the first 12-month proportion will be calculated, based on methods assuming paired samples; in this analysis, each subsequent 12-month proportion would represent comparisons between the first-year proportion and the second-, third-, fourth-, and fifth-year proportions.

An exact upper 95% confidence limit of the difference between the subsequent 12-month proportions (for Years 2, 3, 4, and 5) compared to the first 12-month proportion for patients with data at both year 1 and year k that is less than 20% will reject the null hypothesis in favor of the alternative hypothesis and demonstrate that the proportions are not substantially worse during each of the subsequent evaluation periods.

Final conclusions regarding the durability of effectiveness (beyond 1 year) will be based on completing the 5 year follow-up of all subjects who are still in the study at that time.

A sensitivity analysis (tipping-point analysis) will be performed to assess the impact of patients with inadequate follow-up on the evaluations of the primary endpoint. The tipping-point analysis will be on the primary endpoint using matched pairs and will be performed as follows: assuming no loss to follow-up and given the observed number of patients evaluated at 1 year and k years, for all combinations of success/failure for patients with missing data, the primary endpoint will be evaluated until the point at which the conclusion of the study changes.

#### 2.2 Secondary Endpoints

The secondary endpoints will include the following additional safety endpoints which will be evaluated annually through Year 5 following treatment with the Alair System:

- Rates of Severe exacerbations (exacerbations / subject / year)
- Respiratory adverse events\* (rates of respiratory adverse events, and proportion of subjects with respiratory adverse events)

- Emergency room visits for respiratory symptoms (rates of emergency room visits and proportion of subjects with emergency room visits for respiratory symptoms)
- Hospitalizations for respiratory symptoms (hospitalizations/ subject/ year and the proportion of subjects with hospitalizations for respiratory symptoms)
- Respiratory Serious Adverse Events (detailed narratives will be provided for each event)
- Pre- and post-bronchodilator FEV<sub>1</sub>
- \* A respiratory adverse event is defined as any sign, symptom, illness, clinically significant abnormal laboratory value, or other adverse medical event associated with the "Respiratory System" that appears or worsens in a subject during a clinical study, regardless of whether or not it is considered related to the procedure used as part of the protocol.

#### 2.2.1 Hypotheses

There is no formal hypothesis for the secondary endpoints.

#### 2.2.2 Statistical Methods

Descriptive statistics will be used to summarize the secondary endpoints. For continuous variables, summaries will include the sample size (N), mean, standard deviation, minimum, and maximum. Proportions will be presented with 95% confidence intervals.

#### 3 GENERAL STATISTICAL METHODS

#### 3.1 Analysis Sets

The Intent-to-Treat (ITT) analysis set will consist of all subjects who have been administered at least one BT procedure. The modified Intent-to-Treat (mITT) analysis set will consist of all subjects who have been administered three BT procedures and have primary endpoint data at year 1 and year 2, 3, 4, or 5, as applicable. Analyses based on the ITT analysis set will be considered primary. Analyses based on the mITT analysis set will be considered supportive.

#### 3.2 Control of Systematic Error/Bias

All subjects who have met the inclusion/exclusion criteria and have signed the ICF will be eligible for enrollment in the study. Visual and/or electronic data review will be performed to identify possible data discrepancies. Manual and/or automatic queries will be created in the EDC system and will be issued to the site for appropriate response. Site staff will be responsible for resolving all queries in the database.

#### 3.3 Number of Subjects per Investigative Site

There is no minimum or maximum number of subjects to be enrolled at each center, however, centers in Canada will be limited to 20% of overall enrollment.

#### 4 ADDITIONAL DATA ANALYSES

#### 4.1 Interim Analyses

No formal interim analyses are planned for the PAS2 Study for the purpose of stopping the study early for declaring effectiveness or for futility.

### 4.2 Subgroup Analyses

Inferential analysis of the subset of subjects enrolled at sites in the United States or in Canada may lack the statistical power to demonstrate that the proportions are not substantially worse during each of the subsequent evaluation periods. Descriptive statistics for the point estimates introduced above will be presented for each subset, however, the primary endpoint analysis of the upper 95% confidence limit of the difference between the subsequent 12-month proportions (for Years 2, 3, 4, and 5) compared to the first 12-month proportion will not be required for the subsets.

Descriptive statistics for the subset of subjects enrolled at sites in the United States or in Canada alone will be provided for each of the secondary endpoints, although no conclusions can be drawn from either subset because of the smaller sample sizes.

Subgroup summaries may be performed for subgroups of interest (e.g. sex, age, etc.).

#### 4.3 Justification of Pooling

The clinical study will be conducted under a common protocol for each investigational site with the intention of pooling the data for analysis. Every effort will be made to promote consistency in study execution at each investigational site.

Pooling analyses will be performed to assess the homogeneity of various characteristics and outcomes (e.g. primary endpoint, baseline characteristics, etc.) across investigational sites. If needed, virtual sites will be formed by combining low enrolling investigational sites within geographical region (United States and Canada); low enrolling sites are defined as having <5 subjects. The combining of investigational sites within region will be accomplished by taking the investigational site with the smallest enrollment and combining it with the investigational site with the largest enrollment (of those not enrolling at least 5 subjects).

Consistency will be investigated across country and investigational sites (after combining low enrolling sites), using statistical tests appropriate to the variable and an alpha level of 0.15.

#### 4.4 Multivariable Analyses

Multivariate analyses will be conducted to explore the impact of baseline characteristics on treatment effect, for both the treatment period and the post-treatment period, including changes from year 1 to year 2 through year 5.

#### 4.5 Other Analyses

Demographic data including, but not limited to, age, race, gender and ethnicity, and baseline characteristics including, but not limited to, AQLQ (asthma quality of life questionnaire), maintenance asthma medication doses (see dose conversions in Section 6.5), pre- and post-bronchodilator forced expiratory volume in one second (FEV<sub>1</sub>), prior 12 month history of severe exacerbations (use of systemic corticosteroids (tablets, suspension, or injection) for asthma

symptoms), and emergency room visits and hospitalizations for respiratory symptoms, will be reported for each subject. Procedural characteristics will also be summarized.

Demographic, baseline clinical information, and procedural characteristics will also be provided separately for the subsets of patients enrolled at sites in the United States and sites in Canada.

#### 4.6 Safety Analyses

Adverse events will be reported for the short-term (treatment period) and for the long-term (post-treatment period). The treatment period will be defined as the day of 1st procedure bronchoscopy till 6 weeks (41 days) after the last procedure bronchoscopy. The post-treatment period will begin at the end of the treatment period (i.e. beginning at 6 weeks [42 days] after the last procedure bronchoscopy) for patients who have at least one post-treatment visit (i.e. 6-week visit or later). Patients who do not have a post-treatment visit will not be counted in post-treatment summaries. Annual summaries will be based on a 365-day period beginning at 6 weeks (42 days) after the last procedure bronchoscopy.

Verbatim terms will be classified to preferred terms and system organ classes using the MedDRA dictionary. The preferred terms and system organ classes will then be tabulated by the treatment period and each year of follow-up. All reported adverse events will be summarized by the number of subjects reporting adverse events, system organ class (SOC), preferred term, severity, seriousness, duration, and relationship to procedure. In the summary of MedDRA coded terms, for the preferred terms listed in Table 3, the system organ class will be changed to "Respiratory, thoracic and mediastinal disorders". The reason for the change in SOC is to conservatively report respiratory-related adverse events since the preferred terms in Table 3 represent events that could be related to respiratory function.

Table 3. Preferred Term that will have the system organ class (SOC) changed to "Respiratory, thoracic and mediastinal disorders" for summary tables

| System<br>Organ Class<br>Code | System Organ Class | Preferred<br>Term Code | Preferred Term |
|---|---|---|---|
| 10005329 | Blood and lymphatic system disorders | 10020094 | Hilar lymphadenopathy |
| 10007541 | Cardiac disorders | 10007617 | Cardio-respiratory arrest |
| | General disorders and administration site conditions | 10008469 | Chest discomfort |
| 10018065 | | 10008479 | Chest pain |
| | | 10062501 | Non-cardiac chest pain |
| | Infections and infestations | 10001076 | Acute sinusitis |
| | | 10006451 | Bronchitis |
| | | 10053160 | Bronchitis viral |
| | | 10009137 | Chronic sinusitis |
| 10021881 | | 10022000 | Influenza |
| 10021881 | | 10023874 | Laryngitis |
| | | 10067321 | Laryngitis fungal |
| | | 10024968 | Lower respiratory tract infection |
| | | 10025028 | Lung abscess |
| | | 10028810 | Nasopharyngitis |

| System<br>Organ Class<br>Code | System Organ Class | Preferred<br>Term Code | Preferred Term |
|---|---|---|---|
| | | 10034835 | Pharyngitis |
| | | 10034839 | Pharyngitis streptococcal |
| | | 10035664 | Pneumonia |
| | | 10035728 | Pneumonia pneumococcal |
| | | 10035730 | Pneumonia primary atypical |
| | | 10062352 | Respiratory tract infection |
| | | 10060693 | Respiratory tract infection |
| | | 10000093 | bacterial |
| | | 10039083 | Rhinitis |
| | | 10040753 | Sinusitis |
| | | 10060841 | Sinusitis bacterial |
| | | 10044008 | Tonsillitis |
| | | 10046306 | Upper respiratory tract infection |
| | | 10047473 | Viral pharyngitis |
| | | 10051513 | Viral sinusitis |
| | | 10047482 | Viral upper respiratory tract infection |
| 10022117 | Injury, poisoning and procedural | 10009913 | Collapse of lung |
| 10022117 | complications | 10069363 | Traumatic lung injury |
| 10028395 | Musculoskeletal and connective tissue disorders | 10050819 | Musculoskeletal chest pain |
| 10029104 | Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 10062042 | Lung neoplasm |
| 10029205 | Nervous system disorders | 10034018 | Parosmia |
| 10029203 | There was system disorders | 10040744 | Sinus headache |

In addition to the complete tabulation of adverse events for all subjects enrolled in the study, adverse events will also be tabulated separately for the subsets of subjects enrolled in sites in the United States and the sites in Canada.

#### 4.7 Changes to Planned Analyses

Any changes to the planned statistical analyses made prior to performing the analyses will be documented in an amended statistical analysis plan approved before performing the analyses. Changes from the planned statistical methods after performing the analyses will be documented in the clinical study report along with a reason for the deviation.

#### 5 VALIDATION

All clinical data reports generated per this plan will be validated per 90702587, Global WI: Clinical Data Reporting Validation.

#### 6 PROGRAMMING CONSIDERATIONS

#### 6.1 Statistical Software

Statistical data review will be performed by the sponsor. Statistical analyses will be performed using SAS System software, version 9.2 or later (Copyright © 2000 SAS Institute Inc., SAS Campus Drive, Cary, North Carolina 27513, USA. All rights reserved).

#### 6.2 Format of Output

Results of analysis will be output programmatically to Word documents from SAS with no manual intervention. All output for the final statistical report will be in the form of a Word document containing tables, figures, graphs, and listings, as appropriate.

#### 6.3 Methods for Handling Missing Data

All patients who are enrolled will be eligible for evaluation, regardless of the treatment that ensues. The effect of missing data for the primary endpoint will be evaluated with a sensitivity (tipping-point) analysis (Section 2.1.3). Statistical models that account for censored data will be employed in appropriate circumstances (e.g., for time-to-event outcomes). Outlier values will be evaluated for their validity; all data will be included unless judged to be invalid.

When calculating rates of adverse events, missing and partial dates will be handled as shown below:

| Partial Date Description | Action Taken |
|---|---|
| Entire onset date is missing | The procedure date will be used for the onset |
| | date. |
| The month and the day of the month are | January 1 will be used for the month and day |
| missing but the year is available | of the onset date. However, if the imputed |
| | date falls before the procedure date, then the |
| | procedure date will be used for the onset date. |
| Day is missing, but the month and year | The 1 <sup>st</sup> will be used as the day of the onset |
| are available | date. However, if the imputed date falls |
| | before the procedure date, then the procedure |
| | date will be used for the onset date. |

#### 6.4 Identification of Severe Exacerbations (SE)

- 1. Filter the medication data (MEDS) to keep all courses of oral corticosteroids (CLASS3=OCS) and other medications that are intravenous uses of the same medications identify those by looking for CLASS3='Other Specify' and lowcase(CLSSP) with values: 'intravenous corticosteriod' 'intravenous corticosteroid iv' 'corticosteroid iv'. Note there are spelling mistakes in the entered data.
- 2. Merge the medication data with the AE data by patient and AE related number (RELAENO) on the medication data with AENUM on the AE data.
- 3. Use the onset date and the resolution date of the AE to determine the length of the SE. If an AE has no resolution date, impute the date of the most recent follow-up (scheduled or

- unscheduled) as the resolution date. For partial onset and resolution dates, impute dates as described in Section 6.3.
- 4. When an AE matches with a course of medication, the AE is considered to be an SE, however, when AEs that are SEs occur too close together, the combined AEs are one SE. If the resolution date of one AE selected as an SE is <=6 days before the onset date of another AE that is an SE, then combine the AEs into one SE. There could be more than two AE combined into a single SE.
- 5. SEs are classified in the time period where the onset date of the SE occurs regardless of the duration of the SE.
- 6. For each time period, count the number of SEs for each patient and whether the patient has an SE or not. Two types of summaries will be done for the SEs (also ER visits and hospitalization) to include the following patients: (1) patients with the follow-up visit or later visit for that time period, and (2) patients from (1) and patients with any SE in the time period.

#### **6.5** Medication Dose Conversions

Table 4. Beclomethasone Equivalents

| Drug | <b>Conversion Factor</b> |
|---------------|--------------------------|
| Budesonide | 1.25 |
| Fluticasone | 2 |
| QVAR | 2.5 |
| Mometasone | 2.5 |
| Triamcinolone | 0.5 |
| Flunisolide | 0.5 |
| Ciclesonide | 2.5 |

Table 5. Salmeterol Equivalents

| Drug | <b>Conversion Factor</b> |
|---------------------|--------------------------|
| Formoterol | 100/24 |
| Formoterol Fumarate | 100/24 |

## 7 REVISION HISTORY

| Document<br>Revision Number | Template<br>Number and<br>Version | Section | Change | Reason for Change |
|---|---|---|---|---|
| AA | NA | All | First version | |
| AB | 90702621,<br>AC | All | <ul> <li>Reorganized SAP to match the standard template (90702621)</li> <li>Replaced sections 2-4 from version AA with a protocol summary</li> <li>Changed the primary statistical analysis for the primary endpoint to be paired instead of a two-group test</li> <li>Update the algorithm for identifying severe exacerbations to be more specific</li> <li>Add Table 3 to describe the reassignment of SOCs</li> </ul> | The original SAP was written by a CRO (QST) before BSC took over statistical support for this study; the SAP was rewritten to conform to the current SAP template and to update statistical methods for the primary endpoint. |